CLINICAL TRIAL: NCT01285349
Title: HIV/STI Prevention for Drug-Involved Couples
Acronym: ConnectII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Louisa Gilbert, Associate Research Scientist in the Faculty of Social Work , Adjunct Assistant Professor of Social Work, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AAAA6653
Record Dates: First submitted 2011-01-21; First posted 2011-01-28 (Estimated); Results first posted 2019-01-14 (Actual); Last update posted 2019-01-14 (Actual); Status verified 2018-07

CONDITIONS: Sexually Transmitted Infections
Keywords: HIV, STI, condom use, drug use,
MeSH Terms: conditions — Sexually Transmitted Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Couple-based HIV prevention (Experimental): 7-session couple-based HIV/STI risk reduction intervention (CSTI)
  Interventions: Behavioral: Couple HIV/STI prevention intervention; Behavioral: Couple-based HIV/STI prevention
- Individual HIV/STI Prevention (Active Comparator): 7-session individual HIV/STI intervention comparison condition (ISTI) provided to the index participant alone, which is identical in content to the CSTI.
  Interventions: Behavioral: Individual HIV/STI prevention
- Couple Wellness Promotion (Placebo Comparator): 7-session couple-based stress reduction intervention (CSR) that serves as an attentional control condition.
  Interventions: Behavioral: Couple Wellness Promotion

INTERVENTIONS:
Behavioral: Couple HIV/STI prevention intervention
  Arms: Couple-based HIV prevention
Behavioral: Couple-based HIV/STI prevention
  Arms: Couple-based HIV prevention
Behavioral: Individual HIV/STI prevention
  Arms: Individual HIV/STI Prevention
Behavioral: Couple Wellness Promotion
  Arms: Couple Wellness Promotion

SUMMARY:
This randomized controlled trial is designed to address gaps in couple-based HIV prevention research by focusing exclusively on HIV negative concordant couples where one or both partners are drug-involved. Building on prior couple-based HIV research that resulted in an evidence-based HIV prevention model for couples (Connect), intervention components were modified to address dyadic drug risk reduction and drug-related unsafe sex and a couple-based HIV risk reduction intervention (Connect II) was designed specifically for drug-involved, HIV negative concordant heterosexual couples at risk for HIV/STIs. For this RCT, couples are recruited primarily through street outreach in drug using locations and randomized into one of three arms: (1) couple-based HIV Risk Reduction condition; (2) individual-based HIV Risk Reduction, which delivered the same content as the couple-based condition but was provided to either the male or female drug-using partner alone; or (3) couple-based Wellness Promotion, which served as an attentional control arm. This RCT tests two major hypotheses: (1) whether the HIV risk reduction intervention provided to the couple or an individual partner would be more efficacious in decreasing number of unprotected acts of intercourse and having a lower cumulative incidence of biologically confirmed STIs over the 12-month follow-up period compared to the Wellness promotion control arm and (2) whether the couple-based HIV risk reduction intervention would be more likely to decrease the number of unprotected acts and have a lower cumulative STI incidence compared to the Individual HIV Risk reduction Arm.

DETAILED DESCRIPTION:
Study Design and Population This prospective, blinded randomized controlled trial was conducted between November 2004 and September 2009 in West Harlem, New York City. Participants were recruited through homeless shelters, soup kitchens, syringe exchange programs, street outreach and "word-of-mouth." Most qualified couples came through street outreach. Recruiters informed potential participants about the study, obtained consent to be screened, and screened them for eligibility. People who seemed to be eligible were asked to invite their main sexual partner to participate. A letter to their partner that introduced the study was given to potential participants. Partners interested in participating were screened. If eligible, the recruiter scheduled the couple for baseline data collection. Participants received monetary compensation for completing the baseline assessment and each follow up assessment. The study was approved by the Institutional Review Board of Columbia University. Written informed consent was obtained from all participants prior to enrollment.

Couples were eligible to participate if both were 18 and older and at least one partner was 18-40; (2) both tested HIV negative using Oratest procedures; (3) both identified each other as main, regular partner, boy/girlfriend, spouse, lover; (4) both reported that they have been together for at least 6 months; (5) both intended to remain together for at least one year; (6) at least one partner reported using illicit drugs in the prior 90 days and was seeking or in drug treatment; (7) at least one partner reported having had unprotected intercourse with the other in the prior 90 days. Additionally, at least one partner had to report one or more of the following HIV risk criteria: (1) having had sex with other partners in the prior 90 days; (2) injecting drugs in the prior 90 days; or (3) self-report being diagnosed with an STI in the prior 90 days. Couples were excluded from the study (1) if either partner reported experiencing severe intimate partner violence in the past year by the other partner as assessed by subscales of the Revised Conflict Tactics Scale (Straus, Hamby et al. 1996); (2) if either partner exhibited a severe cognitive or psychiatric impairment assessed during informed consent (3) if either partner did not have sufficient understanding of English and (4) if either partner reported intentions to have a baby in the next year and to relocate beyond a reasonable distance from the study site in the coming year.

Randomization Couples were randomized to the Couple Risk Reduction, Individual Risk Reduction, or the Couple Wellness Promotion conditions at the time of their arrival at their first session (within 10 days from baseline, allowing sufficient time to receive HIV and STI test results). A random number generator was used to assign each couple to one of the three arms with equal probability. The gender of index participant who reported drug use in the past 90 days and seeking or in substance abuse participant was used as a blocking factor to ensure that couples with drug-involved female and male participants were equally balanced across intervention arms. If both partners met above drug involvement criteria eligibility criteria, one partner was randomly selected as the index participant. The Data Coordinator informed the facilitator and couple as to which condition was assigned, entered the treatment assignment into a case report form that contained only the male and female participants' study identification numbers, and then destroyed the assignment card and envelope.

Procedures All three intervention conditions consisted of seven weekly structured 2-hour sessions delivered by female and male facilitators who had at least a bachelor's degree and 2 years of clinical experience in the HIV prevention field. Facilitators completed 40 hours of training and were trained to deliver all three conditions to minimize the threat of facilitator effects. To ensure the fidelity of implementation of all three conditions, facilitators used structured manuals with detailed implementation protocols and were asked to fidelity assessment forms after each session. In addition, facilitators met for weekly 60-minute group supervision to discuss clinical challenges and adherence to the protocol for all three conditions. All intervention sessions were digitally recorded. Recordings and session-specific quality assurance checklists were reviewed to monitor fidelity of implementation of all three conditions and to provide corrective feedback to facilitators.

The Couple-based HIV risk reduction intervention was guided by social cognitive theory (SCT) (Bandura 1992) and a relationship-oriented ecological framework (Bronfenbrenner 1979) which has been described elsewhere (El-Bassel et al., 2001). The core components of the intervention focus on both sexual and drug risk reduction (1) encouraging both partners to disclose and identify mutual drug-related and sexual risks (2) modeling, role-playing and practicing couple communication, negotiation and problem solving skills that both partners may employ together to reduce their drug-related and sexual risks; (3) practicing technical condom use placement skills along with a broader repertoire of pleasurable safer sex activities and syringe disinfection skills and (4) enhancing both couple's motivation to protect each other and set mutual risk reduction goals. Facilitators are trained to validate the relationship's strengths (e.g., commitment, love, trust) and empower the dyad to enact protective behaviors (El-Bassel, 2001, 2005, 2010C). A safe environment is created where sensitive or taboo topics (e.g., outside sexual partners) related to couple's risks may be disclosed and addressed.

The Individual Risk Reduction Intervention covered the same content, skills and sequencing of activities as the Couple Risk Reduction, but was delivered to either or the male or female drug-involved partner in individual sessions by a facilitator of the same gender. In these individual sessions, facilitators are trained to model and role play communication, negotiation and problem-solving skills with participants and encourage them to practice these HIV-related skills and share HIV information with their partners in homework activities.

The Couple Wellness Promotion comparison intervention was designed to control for Hawthorne effects -- to reduce the likelihood that the effects of Connect II risk reduction intervention could be attributed to non-specific features, such as special attention, dosage and couple interaction. Guided by social cognitive theory, the core components of the intervention consist of 7 weekly sessions and employ the same structure as the HIV risk reduction sessions which focus on maintaining a healthy diet promoting physical fitness in daily routines, promoting age appropriate recommendations for screening for common diseases affecting men and women such as cancers, heart disease, diabetes, etc., improving access to health care services by identifying and addressing service barriers and learning stress-reducing exercises.

The participants in all three conditions provided behavioral and biological outcome data at baseline, immediate post intervention IPT, 6- and 12-month post-intervention time points. An Audio Computer Assisted Self-Interview (ACASI) was used to collect self-reported data on drug-related and sexual behavioral outcomes and socio-demographic variables. ACASI provided both audio and video presentation of the questions and response options on a computer enabling participants with low literacy to respond to questions. ACASI was used collect data on self -reported sexual behaviors from participant with their study partners and with all other partners in the prior 90 days, including number of vaginal and anal intercourse acts, number of unprotected vaginal or anal intercourse acts with their study partners and with all other partners, proportion of condom protected acts of vaginal or anal intercourse (e.g. # of times condoms were used during vaginal sex/# of acts of vaginal intercourse), consistent condom use (e.g. used condom100% of time during vaginal sex), and incidence of concurrent sexual partners in the past 90 days at baseline and all follow-ups. The timeline follow-back method was used to enhance recall of sexual behaviors (REF). The primary behavioral outcome was the number of unprotected acts of vaginal intercourse.

Drug risk behavioral outcomes included whether or not and number of times injecting drugs in the past 90 days and number or times sharing syringes, cookers, cotton, or rinse water with another user in the past 90 days. In addition, self-reported data on frequency and type of drug use in the prior 90 days were collected for the following substances: cocaine, crack, heroin, cannabis, and not prescribed sedatives, opiates and stimulants.

To complement self-reports of primary behavioral outcome, we assessed biologically confirmed STI cumulative incidence over the 12-month follow-up period. All participants were asked to provide a self-collected urine specimen after completing the ACASI. Molecular assay of urine specimens for Chlamydia trachomatis and Neisseria gonorrhoeae using. Urine specimens were assayed for Trichomonas vaginalis using. Participants with positive STI test results were referred for single-dose antimicrobial treatment and risk-reduction counseling per CDC recommendations. If either partner tested positive for an STI, both were recommended for treatment. If participants tested positive for any STI at any assessment visit, they were considered an incident STI case for that visit. HIV testing was repeated at the 12-month follow up assessment using Oratest procedures.

Statistical Analysis To assess intervention effects, multilevel mixed-effects models were constructed. . Each observation at the first level of the model represents an individual measurement at one of the three post-treatment time points. Random effect parameters in the model account for dependencies present with each of two types of grouping, couple and time point. Multilevel mixed-effects Poisson regressions were used to estimate effects of the intervention on the number of unprotected acts of intercourse. Effect estimates are reported as incident rate ratios (IRR) and corresponding 95% confidence intervals. Multilevel mixed-effects linear regressions were used for the proportion of protected acts of intercourse; adjusted mean differences and 95% confidence intervals are reported. Multilevel mixed-effects logistic regressions were used to estimate effects on consistent condom use, having concurrent partners, injecting drugs, sharing needles or syringes, and sharing works, cooker, cotton, or rinse water; for these effect estimates odds ratios (OR) and 95% confidence intervals are reported. Due to the low prevalence of STI at baseline and low cumulative incidence over the follow-up period, the biological outcomes were not included in multilevel analysis.

Orthogonal contrast coding was used to test separately for intervention effect (Couple and Individual Risk Reduction jointly vs. Couple Wellness Promotion) and modality effect (Couple Risk Reduction vs. Individual Risk Reduction) within one model. To test for an intervention effect, the coding for Couple Risk Reduction, Individual Risk Reduction and Health Promotion were +1/3, +1/3, and -2/3 respectively. To test for modality effects, the coding for Couple Risk Reduction, Individual Risk Reduction and Health Promotion were+1/2, -1/2 and 0 respectively. All the multilevel models adjusted for the baseline measure of the outcome and gender. The primary analyses used standard intent-to-treat methods in which all available data on all randomized participants were included.

ELIGIBILITY:
Inclusion Criteria:

Couples were eligible to participate if:

* Both were 18 and older and at least one partner was 18-40
* Both tested HIV negative using Oratest procedures
* Both identified each other as main, regular partner, boy/girlfriend, spouse, lover
* Both reported that they have been together for at least 6 months
* Both intended to remain together for at least one year
* At least one partner reported using illicit drugs in the prior 90 days and was seeking or in drug treatment
* At least one partner reported having had unprotected intercourse with the other in the prior 90 days.

Additionally, at least one partner had to report one or more of the following HIV risk criteria:

* Having had sex with other partners in the prior 90 days
* Injecting drugs in the prior 90 days; or
* Self-report being diagnosed with an STI in the prior 90 days.

Exclusion Criteria:

Couples were excluded from the study:

* If either partner reported experiencing severe intimate partner violence in the past year by the other partner as assessed by subscales of the Revised Conflict Tactics Scale
* If either partner exhibited a severe cognitive or psychiatric impairment assessed during informed consent
* If either partner did not have sufficient understanding of English
* If either partner reported intentions to have a baby in the next year and to relocate beyond a reasonable distance from the study site in the coming year.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 564 (Actual)
Dates: Start 2005-11; Primary Completion 2009-10 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Louisa Gilbert, PhD, Principal Investigator — Columbia University
Locations (1):
- Social Intervention Group/Columbia University School of Social Work, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Data from this study is currently available for public use. Requests to use data should be made to the PI, Louisa Gilbert (lg123@columbia.edu)
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data is currently available.
Access Criteria: Please contact PI for sharing access. Data are available for public use.

REFERENCES:
- [Result] El-Bassel N, Gilbert L, Wu E, Witte SS, Chang M, Hill J, Remien RH. Couple-based HIV prevention for low-income drug users from New York City: a randomized controlled trial to reduce dual risks. J Acquir Immune Defic Syndr. 2011 Oct 1;58(2):198-206. doi: 10.1097/QAI.0b013e318229eab1. PMID 21725249

RESULTS

PARTICIPANT FLOW:
Groups:
- Couple Wellness Promotion: 7-session couple-based stress reduction intervention (CSR) that serves as an attentional control condition.
  Couple Wellness Promotion :
- Couple-based HIV Prevention: 7-session couple-based HIV/STI risk reduction intervention (CSTI)
  Couple HIV/STI prevention intervention :
  Couple-based HIV prevention :
- Individual HIV/STI Prevention: 7-session individual HIV/STI intervention comparison condition (ISTI) provided to the index participant alone, which is identical in content to the CSTI.
  Individual HIV/STI prevention :
Period: Overall Study
Arm/Group | Couple Wellness Promotion | Couple-based HIV Prevention | Individual HIV/STI Prevention
Started | 190 | 190 | 184
Completed | 163 | 170 | 157
Not Completed | 27 | 20 | 27
Not completed — Lost to Follow-up | 27 | 20 | 27

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Couple Wellness Promotion | Couple-based HIV Prevention | Individual HIV/STI Prevention | Total
Number analyzed (Participants) | 190 | 190 | 184 | 564
Age, Categorical [Count of Participants; unit: Participants] — The participants in all 3 conditions provided behavioral and biological outcome data at baseline, immediate post-intervention, and at 6-month and 12-month postintervention time points. An audio computer-assisted self-interview (ACASI) was used to collect self-reported data on drug-related and sexual behavioral outcomes and sociodemographic variables.
  Participants
    <=18 years | 0 | 0 | 0 | 0
    Between 18 and 65 years | 190 | 190 | 184 | 564
    >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.0 (6.8) | 36.1 (7.4) | 37.0 (7.2) | 36.5 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 95 | 95 | 92 | 282
  Male | 95 | 95 | 92 | 282
Region of Enrollment [Number; unit: participants]
  United States | 190 | 190 | 184 | 564

OUTCOME MEASURES:

1. Primary Outcome: Number of Unprotected Acts of Intercourse
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: # of unprotected sex acts at 12 months
Groups:
- Couple-Based Wellness Promotion: 7-session couple-based stress reduction intervention (CSR) that serves as an attentional control condition.
  Couple Wellness Promotion :
Arm/Group | Couple-Based Wellness Promotion | Couple-based HIV Prevention | Individual HIV/STI Prevention
Number analyzed (Participants) | 163 | 170 | 163
# of unprotected sex acts at 12 months | 19.7 (28.1) | 12.9 (19.2) | 18.2 (27.0)

2. Secondary Outcome: Number of Participants With Biologically Confirmed STIs (i.e., Chlamydia, Gonorrhea, and Trichomoniasis)
Time Frame: past 12 months
Measure: Number; unit: participants
Arm/Group | Couple Wellness Promotion | Couple-based HIV Prevention | Individual HIV/STI Prevention
Number analyzed (Participants) | 163 | 170 | 184
participants | 3 | 3 | 2

ADVERSE EVENTS:
Arm/Group | Couple Wellness Promotion | Couple-based HIV Prevention | Individual HIV/STI Prevention
All-Cause Mortality (participants affected / at risk) | 0/190 | 0/190 | 0/183
Serious Adverse Events (participants affected / at risk) | 0/190 | 0/190 | 0/183
Other Adverse Events (participants affected / at risk) | 0/190 | 0/190 | 0/183

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes